CLINICAL TRIAL: NCT02867007
Title: Multicenter, Open-label, Phase 1, Dose-escalation, Cohort-expansion, First-in-Human Study of KHK2455 Administered as Monotherapy and in Combination With Mogamulizumab in Adult Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: KHK2455 Alone and in Combination With Mogamulizumab in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2455-001
Expanded Access: NCT04321694 (No longer available)
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor; Cancer; Carcinoma
Keywords: KW-0761; KHK2455; Metastatic Solid Tumors; Locally Advanced Solid Tumors; Mogamulizumab; Oncology; Anti-Tumor
MeSH Terms: conditions — Neoplasms; Carcinoma | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KHK2455 + Mogamulizumab (Experimental): Part 1 (Dose Escalation Part): Will identify the MTD for the KHK2455 monotherapy run-in and for the combination regimen (KHK2455 monotherapy [Cycle 0] followed by KHK2455 +mogamulizumab combination [Cycle 1]).
  Part 2 (Expansion Part): Subjects with a selected tumor type will be enrolled and treated with the recommended dose of KHK2455 established in Part 1 in combination with mogamulizumab.
  Interventions: Drug: KHK2455; Drug: Mogamulizumab

INTERVENTIONS:
Drug: KHK2455 — oral dosing
Drug: Mogamulizumab — i.v. administration
  Other Names: Mogamulizumab: KW-0761; Poteligio

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, and determine the maximum tolerated dose (MTD) or the highest protocol-defined dose, in the absence of exceeding the MTD, of KHK2455 administered orally in combination with mogamulizumab to subjects with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The study is designed as a 2-part, multicenter, open-label, Phase 1, dose-escalation, cohort-expansion study of KHK2455 as a monotherapy run-in (Cycle 0) followed by combination therapy with the anti-CCR4 antibody mogamulizumab (Cycle 1 and beyond).

Part 1 will identify the MTD or the highest protocol-defined dose, in the absence of exceeding the MTD, for the KHK2455 monotherapy run-in and for the combination regimen (KHK2455 monotherapy [Cycle 0] followed by KHK2455 + mogamulizumab combination [Cycle 1]). The dose escalation phase (Part 1) will enroll up to approximately 36 subjects.

Part 2, the cohort-expansion phase, will further explore the safety, tolerability, PK, PD, pharmacogenomics (PGx), and preliminary anti-tumor activity of KHK2455 administered as monotherapy and in combination with mogamulizumab in subjects with one cohort-specific tumor type. In Part 2, approximately 15 subjects with a selected tumor type will be enrolled and treated with the recommended KHK2455 dose established in Part 1 in combination with mogamulizumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have histological or cytological evidence of a solid malignancy
* Subject must have measurable neoplastic disease according to the RECIST v1.1;
* Subject must have locally advanced or metastatic solid tumor with no additional therapy options available that are known to provide clinical benefit per institutional standards;
* Subject is able to understand and willing to sign the ICF, according to institutional standards, prior to the initiation of any study related procedures;
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Subject must have a life expectancy of > 3 months, in the Investigator's judgment;
* Subject must have a left ventricular ejection fraction of ≥ 50%;
* Subject must have adequate organ function as defined below. The following parameters must be evaluated within 28 days prior to Cycle 0 Day 1 (monotherapy run-in period):

  * Aspartate aminotransferase (AST) and/or ALT ≤ 2.5 × ULN
  * Total bilirubin ≤ 1.5 × ULN
  * Hemoglobin ≥ 9.6 g/dL
  * Serum creatinine ≤ 2.0 × ULN
  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm3
  * Absolute lymphocytes count ≥ 800 cells/mm3
  * Platelets ≥ 100 × 109/L
  * Albumin ≥ 2.0 g/dL
* Subject has recovered (i.e., to Grade ≤ 1 or to a baseline level) from the effects of surgery, radiotherapy, chemotherapy, hormonal therapy, or other therapies for cancer; with the exception of vitiligo, alopecia, neuropathy, partial hearing loss, and/or endocrinopathies (for which no resolution is required);
* Subject on prior chemotherapeutic, immunomodulator (such as anti-CTLA-4, anti-PD-1 or anti-PD-L1 inhibitor), investigational, or other therapies for the treatment of cancer must wait at least 28 days after the last dose of these therapies before administration of the first dose of the IMP.
* Male subject and woman of child-bearing potential (WOCBP) must agree to use a medically-effective, double-barrier method of contraception (as defined in the ICF) to prevent pregnancy while on study and for 6 months after the last dose of IMP. WOCBP includes any female who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea ≥ 12 consecutive months without an alternative medical cause). If the subject is a WOCBP, she must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Cycle 0 Day 1 (monotherapy run-in period; prior to receiving KHK2455);
* Subject must have a brain scan performed during Screening or within 3 months prior to signing informed consent;
* Subject must be able to swallow solid dosage forms.

Exclusion Criteria:

* Subject is enrolled (concurrently) in another investigational study, with the exception of the follow-up period of another investigational study in which no anti-cancer therapy is being administered and where only data are being collected;
* Subject who has been previously treated with an anti-CCR4 antibody or an IDO1 inhibitor;
* Subject with a history of severe hypersensitivity reactions to any of the other excipients of the protocol IMPs (see Section 8.1.1);
* Subject is a female who is pregnant or breast-feeding, or intends to become pregnant during their participation in the study (including up to 6 months after the last dose of IMP) or is a male who intends to father a child during their participation in the study (including up to 6 months after the last dose of IMP);
* Subject has known primary immunodeficiency or active tuberculosis or tests positive for acquired human immunodeficiency virus;
* Subject who tests positive for hepatitis B surface antigen (HBVsAg) or hepatitis C ribonucleic acid (RNA) indicating acute or chronic infection;
* Subject who has undergone a major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of KHK2455 or is still recovering from prior surgery;
* Subject has a mean QT interval corrected for heart rate using Bazett's (QTcB) or Fridericia's (QTcF) correction ≥ 500 ms calculated from 3 consecutive 12-lead ECGs at Screening;
* Subject with an uncontrolled concurrent illness including, but not limited to, ongoing or active infection, significant hepatic disease (subjects with liver metastases who meet the inclusion criteria will be allowed ), pneumonitis, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial or other current severe lung disease including poorly controlled chronic obstructive pulmonary disease, malabsorption or protracted diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent;
* Subjects with Gilbert's syndrome;
* Subject with known active CNS metastasis, except primary brain tumors. Subjects with asymptomatic brain metastases or spinal cord compression who have been treated, are considered stable, and have not received steroid doses > 10 mg/day of prednisolone equivalent to treat these conditions prior to consent may be included;
* Subject with any prior Grade ≥ 3 irAE to other therapeutic proteins or immunotherapy, and the reaction could not be controlled or prevented on subsequent infusion with standard therapies such as antihistamines, 5-hydroxytryptamine antagonists, or corticosteroids;
* Subject with a history of organ transplant or allogeneic bone marrow transplant;
* Subject currently using or have received immunosuppressive medications within 14 days prior to the first dose of KHK2455, with the exception of topical or systemic corticosteroids that are not to exceed 10 mg/day of prednisone or equivalent;
* Subject with a history of autoimmune disease (e.g., ulcerative colitis, Crohn's disease, rheumatoid arthritis, Addison's syndrome, multiple sclerosis, uveitis, systemic lupus erythematosus or Wegener's granulomatosis). Subjects with vitiligo, endocrinopathies, and alopecia are allowed. Subjects with psoriasis not requiring systemic treatment within the past 6 months are allowed;
* Subject who has a history of second primary cancer within the past 5 years, with the exception of:

  * Curatively resected non-melanoma skin cancer;
  * Curatively treated cervical intraepithelial neoplasia or prostate carcinoma with current prostate specific antigen < 0.01 ng/mL; or
  * Curatively treated ductal carcinoma in situ of the breast.
* The subject has a condition(s) that, in the opinion of the Investigator and/or Sponsor, would interfere with evaluation of the IMP or interpretation of the subject's safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08; Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 2 years
  Safety assessment variables will include all adverse events (AEs) including serious and non-serious AEs, changes in clinical laboratory parameters, vital signs, 12-lead electrocardiograms, physical examination, and immunogenicity

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Tampa, Florida
  - Albuquerque, New Mexico
  - Houston, Texas
- Paris, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yap TA, Rixe O, Baldini C, Brown-Glaberman U, Efuni S, Hong DS, Massard C, Muzaffar J, Varga A, Yilmaz E, Ikawa Y, Shiue LH, Liu Y, Hruska MW, Zhao H, Tokunaga A, Sahebjam S. First-in-human phase 1 study of KHK2455 monotherapy and in combination with mogamulizumab in patients with advanced solid tumors. Cancer. 2025 Jul 1;131(13):e35939. doi: 10.1002/cncr.35939. PMID 40536766